CLINICAL TRIAL: NCT05282381
Title: Decisional Regret in a Prospective Cohort of Renal Transplant Recipients: the DONOR Study
Brief Title: Evaluation of Regret in Kidney Transplantation
Acronym: DONOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0272; 2021-A02002-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Renal Transplant Candidate for Right Kidney; Renal Transplant Candidate for Left Kidney
Keywords: Decisional regret; Kidney transplantation; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of renal transplant recipients
  Interventions: Behavioral: DRS : Decision Regret Scale

INTERVENTIONS:
Behavioral: DRS : Decision Regret Scale — The DRS is a self-administered questionnaire including 5 items assessing decisional regret in a score graduated between 0 and 100 (0 = no regret).This scale is associated with the ReTransQoL, a specific quality of life questionnaire.
  Questionnaires are administrated at 1, 3, 6 and 12 months post-transplantation.

SUMMARY:
Decisional regret is a negative feeling, involving distress or remorse following a decision. This has been studied in several areas such as psychology, economy or marketing. Patients suffering from end-stage renal disease may choose between dialysis and transplantation. This decision-making process is shared with the nephrologist, who explained to the patient the pros and cons of these two possibilities. Although transplantation offers a better life expectancy and quality of life than dialysis, nothing is known about the proportion of patients regretting their choice to be transplanted. The DONOR study aims to determine the proportion of patients regretting their decision, in a prospective cohort of renal transplant recipients. The decisional regret will be assessed by the DRS ("Decisional Regret Scale"), associated with the RetransQoL, a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation in the Lille University Hospital
* Functional kidney graft after 28 days post transplantation

Exclusion Criteria:

* Previous other solid organ transplant
* Combined transplantation (kidney and liver for example)
* Cognitive disorders
* Lack of French language skill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a kidney transplant in the nephrology department of the Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Decisional regret at 12 months post kidney transplantation, defined as a score ≥30 on the Decisional Regret Scale | At 12 months post-transplantation
  The decisional regret scale consists of five items addressing the notion of regret from different perspectives. The patient is asked to respond to each item using a 5-point Likert-type scale. The results of the Decisional Regret Scale are converted into a score from 0 to 100, with values increasing in multiples of 5. A score of 0 means no regret.
  Three categories of the DRE score were created: no regret (score = 0), low regret (score between 5 and 25), and moderate to high regret (score ≥ 30

SECONDARY OUTCOMES:
Specific Quality of Life Scale (ReTransQoL) | At 1, 3, 6 and 12 months post-transplantation
  The ReTransQoL (Renal Transplant Quality of Life) questionnaire is a quality of life related-questionnaire, specific for kidney transplant recipients and developed by Gentile et al. in 2008 (Gentile et al, Health Qual Life Outcomes, 2008). It consists in 49 items, divided into 5 dimensions: Physical Health, Medical Care, Fear of losing the Graft, Treatment and Mental Health. This results in a quality of life score, from 0 to 100 (0 being the lowest quality of life score).
Variation of decisional regret over time, following kidney transplantation, using the Decisional Regret Scale | At 1, 3, 6 and 12 months post-transplantation
  The decisional regret scale consists of five items addressing the notion of regret from different perspectives. The patient is asked to respond to each item using a 5-point Likert-type scale. The results of the Decisional Regret Scale are converted into a score from 0 to 100, with values increasing in multiples of 5. A score of 0 means no regret.
  Three categories of the DRE score were created: no regret (score = 0), low regret (score between 5 and 25), and moderate to high regret (score ≥ 30
Identification of biological, psychological and sociological risk factors for decisional regret at 12 months post kidney transplantation, defined as a score ≥30 on the Decisional Regret Scale | At baseline, and during the 12 months follow-up period.
  The decisional regret scale consists of five items addressing the notion of regret from different perspectives. The patient is asked to respond to each item using a 5-point Likert-type scale. The results of the Decisional Regret Scale are converted into a score from 0 to 100, with values increasing in multiples of 5. A score of 0 means no regret.
  Three categories of the DRE score were created: no regret (score = 0), low regret (score between 5 and 25), and moderate to high regret (score ≥ 30

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Maanaoui, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France